CLINICAL TRIAL: NCT00389103
Title: A Phase 1, Placebo-Controlled, Double-Blind Study of the Safety and Immunogenicity of Two Injections of MVA3000 Modified Vaccinia Ankara (MVA) Smallpox Vaccine in Vaccinia Naive Adult Subjects With a History of Atopic Dermatitis (AD)
Brief Title: Safety Study of MVA Smallpox Vaccine in Subjects With a History of Atopic Dermatitis (AD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Senior management decision
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-249-005
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Smallpox; Atopic Dermatitis
MeSH Terms: conditions — Smallpox; Dermatitis, Atopic | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- placebo (Placebo Comparator)
  Interventions: Biological: MVA (smallpox vaccine)

INTERVENTIONS:
Biological: MVA (smallpox vaccine) — 0.5ml of MVA3000 Smallpox vaccine, administered twice separated by 28 days, subcutaneous injections
  Other Names: placebo

SUMMARY:
purpose of this study is to assess the safety and immunogenicity of two MVA smallpox vaccine injections in healthy adults that are 18-35 years of age with a history of mild to moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. subjects will be randomized to receive investigational vaccine or placebo at a ratio of 3.5:1, MVA3000 to placebo. All subjects will undergo a screening period, a treatment/observation period during which all subjects will receive injections on study day 0 and study day 28 of investigational vaccine or placebo. The clinical observation period will be completed at day 56. A visit will occur at approximately 3 months after the second study injection (study day 118) for additional blood collection and a review of the subject's health status. Follow-up will be obtained via telephone contacts approximately 6 months after the end of the second injection during the treatment/observation period.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old and who were born after 1971 with no previous history of smallpox vaccination
* Subjects must be in good general health Female subjects must not be pregnant or lactating and must agree to practice birth control during the course of the study
* Subjects must have a diagnosis of AD by an experienced clinician that includes a history of both major and minor diagnostic criteria
* At the time of screening, the subject must have "mild to moderate" AD.

Exclusion Criteria:

* History or evidence of prior exposure to a vaccinia or MVA- containing product
* known or suspected history of immunodeficiency other than AD
* Known or suspected impairment of major organ function
* Known history or diagnosis of cardiac disease or cerebrovascular disease
* presence of acute, chronic, or active exfoliative skin conditions other than AD, open wounds, or burns.
* Dementia or history of seizures
* Known allergies to MVA or any known components of the vaccine
* transfusion of blood, organ transplantation, or treatment with any blood product
* morbid obesity, or a BMI less than or equal to 18.5
* history of or current drug or alcohol abuse (except nicotine) within the past 6 months or any history of IV drug use
* history of major psychiatric illness except major depression not requiring medical therapy.
* subjects who have participated in another investigational drug or vaccine trial within 30 days of study day 0

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety | Study Completion

SECONDARY OUTCOMES:
Immunogenicity | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (3):
- United States (3):
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Oregon Health & Science University, Portland, Oregon
  - DermResearch, Inc., Austin, Texas

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com